CLINICAL TRIAL: NCT02410174
Title: Phase I Trial of Stereotactic Body Radiotherapy (SBRT) of the Primary Tumor in Renal Cell Carcinoma (RCC)
Brief Title: To Evaluate Stereotactic Body Radiotherapy for Treatment of Primary Renal Cell Carcinoma Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Poor Accural
Sponsor: Beth Israel Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 100-11
Record Dates: First submitted 2015-04-02; First posted 2015-04-07 (Estimated); Last update posted 2017-01-09 (Estimated); Status verified 2016-04

CONDITIONS: Primary Tumor; Renal Cell Carcinoma
Keywords: Renal Cell Carcinoma; RCC; Stereotactic Body Radiotherapy; SBRT
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Stereotactic Body Radiotherapy (SBRT) (Experimental): Starting dose of 48Gy in 3 fractions, will escalate dose by 2 Gy per fraction (a 6Gy total dose) to a maximum dose of 20Gy x 3 fractions (TD 60 Gy in 3 fractions).
  Interventions: Radiation: Stereotactic Body Radiotherapy (SBRT)

INTERVENTIONS:
Radiation: Stereotactic Body Radiotherapy (SBRT)

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of the use of stereotactic body radiotherapy (SBRT) for the treatment of the primary tumor in renal cell carcinoma (RCC) in medically inoperable patients and/or patients who refuse surgery. Standard treatment of RCC is surgery. A number of non-surgical treatments of RCC are also available, but are highly invasive and are associated with significant side effects. SBRT is a non-invasive, non-surgical treatment that requires tumor immobilization and image guidance in order to deliver a very precise, high-dose treatment. This trial will assess the use of SBRT to treat primary renal tumors by determining the maximum tolerated dose and toxicity. Subjects enrolled in this study will then be followed and evaluated for toxicity, serum chemistry, complete blood count, and urinalysis. In addition, they will undergo renal scans to assess the functionality of their renal tissue.

DETAILED DESCRIPTION:
There is a need for a non-invasive treatment modality in renal cell carcinoma (RCC) patients who are medically or technically inoperable or refuse surgery. The primary tumor in patients with RCC is generally managed surgically or with a non-surgical ablative modality, but there is significant toxicity and invasiveness associated with current surgical and percutaneous treatment modalities. Stereotactic radiotherapy was first developed to treat brain metastases and other intracranial tumors by giving a single high-dose treatment delivered with a precision of less than 1 mm. This treatment requires immobilization of the tumor and precise imaging to guide the treatment. The brain is particularly amenable to this approach since there is no internal brain motion, the skull is easily fixed in position, and excellent imaging is available. Recent developments in immobilization and image guidance now permit precise tumor targeting of extracranial sites, such as the liver and lung. Stereotactic radiotherapy used at extracranial sites is called stereotactic body radiotherapy (SBRT). Because of the great precision of SBRT, a high dose per treatment is possible. Early work evaluating SBRT in primary and metastatic liver and lung tumors has shown excellent results in tumor control and toxicity. Based on this, we propose expanding the use of this technique to RCC.

In this study, the investigators seek to evaluate the safety and efficacy of SBRT for the treatment of the primary tumor in renal cell carcinoma (RCC). One goal of this study is to establish the maximum tolerated dose (MTD) of renal SBRT by determining the dose-volume relationship and toxicity for the kidney when high dose per fraction SBRT is used. In order to ensure proper immobilization and tumor localization, the investigators will use abdominal compression, 4D CT scanning at the time of simulation, and cone beam CT scanning at the time of treatment. The investigators propose to perform Tc-99m glucoheptonate renal scans before and after SBRT to assess renal tissue at the periphery of the lesion, as well as baseline and follow-up serum chemistry evaluation, creatinine, complete blood count, urinalysis, and creatinine clearance.

ELIGIBILITY:
Inclusion Criteria:

* Any patient with a primary renal cell carcinoma (RCC) tumor who is inoperable for technical (i.e surgical) or medical reasons
* Patient must be screened by a urologic surgeon to verify eligibility on the above basis
* Biopsy proof of RCC is preferred; however, in current practice the diagnosis is often clinical based on characteristic imaging. If there are compelling clinical reasons not to proceed with biopsy, the clinical diagnosis will suffice.
* Patient with metastases are eligible if in the opinion of the treating physicians the patient could benefit from treatment of the primary renal tumor.
* ECOG performance status 0-2
* Age ≥18 years
* Signed informed consent

Exclusion Criteria:

* Inadequate renal function, as measured by creatinine clearance calculated from 24 hour urine collection. Creatinine clearance values of at least 50 ml/min are required
* Prior attempt at curative treatment of this primary kidney tumor
* Inability to lie still for approximately 1 hour in immobilization device
* Presence of a connective tissue disorder other than rheumatoid arthritis.
* Pregnancy
* Inability to develop a radiation treatment plan that adheres to the dose constraints described below in Radiotherapy Treatment Planning section.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2012-05; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Local Failure | up to 10 years
  A ≥20% increase in the sum of the diameters of the tumor with a minimum increase in the sum of 5 mm (RECIST criteria) or any areas of enhancement on follow up imaging studies is categorized as progression. Time to failure will be from the last date of SBRT to date of local failure or last follow-up.
  * Local failure will be classified as in field if it occurs within the treated volume or marginal if it occurs at the edge of the treated volume.
  * Development of a new renal tumor elsewhere in the kidney. This will not be considered a local failure. Time to development of a new tumor elsewhere in the kidney will be from the last date of SBRT to date of the event or last follow-up.

SECONDARY OUTCOMES:
Regional Nodal Failure | up to 10 years
  -Recurrence is renal hilar, para-aortic or para-caval lymph nodes.
Metastases | up to 10 years
  Incidence of metastases
Overall survival | up to 10 years
Serum Creatinine Level | 1 year
24 Hour Creatinine Clearance | 1 year
Results of Tc-99m Glucoheptonate Renal Scan | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Ronald D Ennis, MD, Principal Investigator — Mount Sinai Beth Israel
Locations (2):
- United States (2):
  - Mount Sinai Beth Israel Hospital, New York, New York
  - Mount Sinai Roosevelt Hospital, New York, New York